CLINICAL TRIAL: NCT05564052
Title: A Randomized, Controlled, Open-label, Multicenter, Inferentially Seamless Phase 2/3 Study of Ibrutinib in Combination With Rituximab Versus Physician's Choice of Lenalidomide Plus Rituximab or Bortezomib Plus Rituximab in Participants With Relapsed or Refractory Mantle Cell Lymphoma
Brief Title: A Study of Ibrutinib With Rituximab in Relapsed or Refractory Mantle Cell Lymphoma
Acronym: VEGA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109252; 54179060MCL3004 (Other: Janssen Research & Development, LLC); 2022-000364-21 (EudraCT Number); 2023-503618-64-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2022-09-30; First posted 2022-10-03 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Lymphoma, Mantle-Cell
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — ibrutinib; Lenalidomide; Rituximab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 2: Treatment Arm A1 (Rituximab plus Ibrutinib) (Experimental): Participants will receive rituximab 375 milligrams per meter square (mg/m^2) intravenously (IV) on Day 1 of Cycles 1 to 6 with ibrutinib 560 milligrams (mg) orally, once daily starting on Day 1 of Cycle 1 until disease progression or unacceptable toxicity (each cycle length is 28 days).
  Interventions: Drug: Ibrutinib; Drug: Rituximab
- Phase 2: Treatment Arm A2 (Rituximab plus Ibrutinib) (Experimental): Participants will receive rituximab 375 mg/m^2 IV on Day 1 of Cycles 1 to 6 with ibrutinib 420 mg orally, once daily starting on Day 1 of Cycle 1 until disease progression or unacceptable toxicity (each cycle length is 28 days).
  Interventions: Drug: Ibrutinib; Drug: Rituximab
- Phase 2: Treatment Arm A3 (Rituximab plus Ibrutinib) (Experimental): Participants will receive rituximab 375 mg/m^2 IV on Day 1 of Cycles 1 to 6 with ibrutinib 140 mg orally, twice daily starting on Day 1 of Cycle 1 until disease progression or unacceptable toxicity (each cycle length is 28 days).
  Interventions: Drug: Ibrutinib; Drug: Rituximab
- Phase 2: Treatment Arm B (Rituximab plus Lenalidomide or Bortezomib) (Experimental): Participants will receive rituximab 375 mg/m^2 IV on Day 1 of Cycles 1 to 6 (each cycle length is 21 or 28 days) with physician's choice of either lenalidomide 20 mg orally, once daily from Day 1 through Day 21 of 28-day cycle or bortezomib 1.3 mg/m^2 IV or subcutaneously (SC) on Days 1, 4, 8 and 11 of a 21-day cycle until disease progression or unacceptable toxicity.
  Interventions: Drug: Lenalidomide; Drug: Rituximab; Drug: Bortezomib

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib capsules will be administered orally.
  Other Names: JNJ-54179060, IMBRUVICA, PCI-32765
  Arms: Phase 2: Treatment Arm A1 (Rituximab plus Ibrutinib); Phase 2: Treatment Arm A2 (Rituximab plus Ibrutinib); Phase 2: Treatment Arm A3 (Rituximab plus Ibrutinib)
Drug: Lenalidomide — Lenalidomide capsules will be administered orally.
  Arms: Phase 2: Treatment Arm B (Rituximab plus Lenalidomide or Bortezomib)
Drug: Rituximab — Rituximab will be administered IV.
Drug: Bortezomib — Bortezomib will be administered either intravenously or subcutaneously.
  Arms: Phase 2: Treatment Arm B (Rituximab plus Lenalidomide or Bortezomib)

SUMMARY:
The purpose of this study is to provide continued access to treatment for participants who continue to benefit from treatment.

DETAILED DESCRIPTION:
Mantle cell lymphoma (MCL) is an uncommon and incurable clinicopathologic subtype of B-cell non-Hodgkin Lymphoma (NHL). Ibrutinib is a first-in-class potent, orally administered, covalently-binding small molecule inhibitor of Bruton's tyrosine kinase (BTKi) for the treatment of B-cell malignancies and chronic graft-versus-host disease. The primary hypothesis of the study is to provide continued access to treatment for participants who continue to benefit from treatment. The study will include a screening phase (up to 30 days prior to randomization), a treatment phase (from randomization until study treatment discontinuation). safety assessments include adverse events (AEs), serious adverse events (SAEs), clinical laboratory tests, vital signs, electrocardiogram (ECG), physical examination. The Phase 2 exploratory objectives and endpoints of characterization of pharmacokinetic and pharmacodynamic of ibrutinib may continue to be evaluated using blood samples already collected. The total duration of the study will be up to 2 years 1 month.

ELIGIBILITY:
Inclusion Criteria:

* At least 1 prior treatment regimen for mantle cell lymphoma (MCL) excluding inhibitor of Bruton's tyrosine kinase (BTKi)
* Documented disease progression or relapse following the last anti-MCL treatment
* At least 1 measurable site of disease on cross-sectional imaging that is greater than or equal to (>=) 2.0 centimeters (cm) in the longest diameter and measurable in 2 perpendicular dimensions per computed tomography (CT)
* Eastern Cooperative Oncology Group (ECOG) performance status score 0 or 1

Exclusion Criteria:

* Prior therapy with ibrutinib or other BTK inhibitor
* Prior treatment with both lenalidomide and bortezomib. Prior treatment with only 1 of these therapies is allowed
* Major surgery within 4 weeks of randomization
* Concurrent enrollment in another therapeutic investigational study
* Known central nervous system lymphoma
* History of stroke or intracranial hemorrhage within 6 months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-12-06 (Actual); Primary Completion 2023-12-06 (Actual); Study Completion 2024-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (66):
- Brazil (11):
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte
  - Sociedade Beneficente de Senhoras - Hospital Sirio Libanes HSL Unidade Brasilia, Brasília
  - Ynova Pesquisa Clinica, Florianópolis
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Complexo Hospitalar de Niteroi, Niterói
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital Das Clinicas Da Faculdade De Medicina De RPUSP HCRP, Ribeirão Preto
  - Oncoclinicas Rio de Janeiro S A, Rio de Janeiro
  - Instituto de Ensino e Pesquisa Sao Lucas - IEP HEMOMED, São Paulo
  - Instituto D Or de Pesquisa e Ensino IDOR, São Paulo
  - Casa de Saude Santa Marcelina - Hospital Santa Marcelina, São Paulo
- Czechia (3):
  - Fakultni Nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Kralovske Vinohrady, Prague
  - General University Hospital in Prague, Prague
- Greece (3):
  - Attikon University General Hospital of Attica, Athens
  - University Hospital of Ioannina, Ioannina
  - G.Papanikolaou, Thessaloniki
- India (8):
  - Healthcare Global (HCG) Hospital, Bangalore
  - American Oncology Institute Cancer Treatment Hospital Hyderabad, Hyderabad
  - Bhagwan Mahaveer Cancer Hospital & Research Centre, Jaipur
  - HCG cancer center, Jaipur
  - Tata Medical Center, Kolkata
  - AMRI Hospital, Mukundapur, Mukundapur
  - Deenanath Mangeshkar Hospital and Research Centre, Pune
  - Synergy Superspeciality Hospital, Rajkot
- Malaysia (5):
  - Hospital Ampang, Ampang
  - Hospital Sultanah Aminah, Johor Bharu
  - Hospital Queen Elizabeth, Kota Kinabalu
  - University Malaya Medical Centre, Kuala Lumpur
  - Subang Jaya Medical Centre, Subang Jaya
- Poland (9):
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im Ks B Markiewicza, Brzozów
  - Swietokrzyskie Centrum Onkologii SPZOZ w Kielcach, Kielce
  - Uniwersytecki Szpital Kliniczny Nr 1 w Lublinie, Lublin
  - Szpital Specjalistyczny im Jedrzeja Sniadeckiego w Nowym Saczu, Nowy Sącz
  - SPZOZ Ministerstwa Spraw Wewnetrznych z Warminsko Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
  - Centrum Medyczne Pratia Poznan, Skorzewo
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 PUM im prof Tadeusza Sokolowskiego w Szczecinie, Szczecin
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
  - Specjalistyczny Szpital im dra Alfreda Sokolowskiego w Walbrzychu, Wałbrzych
- Auxilio Mutuo Cancer Center, San Juan, Puerto Rico
- Romania (2):
  - Spitalul Clinic Coltea, Bucharest
  - Ovidius Clinical Hospital OCH, Ovidiu
- Spain (5):
  - Hosp Reina Sofia, Córdoba
  - Hosp. Univ. Infanta Leonor, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp Clinico Univ de Salamanca, Salamanca
- Sweden (2):
  - Falu Lasarett Medicinkliniken Falun, Falun
  - Sunderby Sjukhus, Luleå
- Taiwan (4):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Chi Mei Medical Center Liu Ying, Tainan
  - National Taiwan University Hospital, Taipei
- Thailand (6):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao Hospital and Medical College, Bangkok
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Maharaj Nakorn Chiang Mai hospital Faculty of Medicine, Chiang Mai
  - Srinagarind Hospital, Khon Kaen
- Turkey (Türkiye) (7):
  - Ankara Bilkent Sehir Hastanesi, Ankara Sehir Hastanesi
  - Ondokuz Mayis University, Atakum
  - Trakya University Medical Faculty, Edirne
  - Medipol Mega University Hospital, Istanbul
  - Istanbul University, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
  - Sakarya Egitim Ve Arastırma Hastanesi Korucuk Kampus, Sakarya

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was planned to be conducted in 2 parts: Phase 2 and Phase 3. However, due to early termination of enrollment, no participants were enrolled on the Phase 3 part of the study. Hence, the results were only presented for Phase 2 part. Participants with relapsed or refractory mantle cell lymphoma were enrolled in the study.
Groups:
- Arm A1: Ibrutinib 560 mg + Rituximab 375 mg/m^2: Participants received ibrutinib 560 milligrams (mg; 4 capsules of 140 mg) orally once daily (QD) in each 28-day treatment cycle starting from Cycle 1 Day 1 until disease progression or unacceptable toxicity. Participants also received rituximab 375 milligrams per meter square (mg/m^2) intravenous (IV) infusion on Day 1 of each 28-day treatment cycle from Cycles 1 to 6. After implementation of Protocol Amendment 1 (dated 08 June 2023), all participants were given the option either to continue with the randomized treatment arm or switch to ibrutinib monotherapy to receive ibrutinib 560 mg capsules orally QD (unless the dose was previously reduced) until the investigator determined that the participant was no longer benefiting from treatment (disease progression or unacceptable toxicity had occurred), the participant withdrew consent, alternative access to study treatment was available and feasible, or until the end of the study, whichever occurred earlier.
- Arm A2: Ibrutinib 420 mg + Rituximab 375 mg/m^2: Participants received ibrutinib 420 mg (3 capsules of 140 mg) orally QD in each 28-day treatment cycle starting from Cycle 1 Day 1 until disease progression or unacceptable toxicity. Participants also received rituximab 375 mg/m^2 IV infusion on Day 1 of each 28-day treatment cycle from Cycles 1 to 6. After implementation of Protocol Amendment 1 (dated 08 June 2023), all participants were given the option either to continue with the randomized treatment arm or switch to ibrutinib monotherapy to receive ibrutinib 560 mg capsules orally QD (unless the dose was previously reduced) until the investigator determined that the participant was no longer benefiting from treatment (disease progression or unacceptable toxicity had occurred), the participant withdrew consent, alternative access to study treatment was available and feasible, or until the end of the study, whichever occurred earlier.
- Arm A3: Ibrutinib 140 mg + Rituximab 375 mg/m^2: Participants received ibrutinib 140mg (1 capsule of 140mg) orally twice daily (BID) in each 28-day treatment cycle starting from Cycle 1 Day 1 until disease progression or unacceptable toxicity. Participants also received rituximab 375 mg/m^2 IV infusion on Day 1 of each 28-day treatment cycle from Cycles 1 to 6. After implementation of Protocol Amendment 1 (dated 08 June 2023), all participants were given the option either to continue with the randomized treatment arm or switch to ibrutinib monotherapy to receive ibrutinib 560 mg capsules orally QD (unless the dose was previously reduced) until the investigator determined that the participant was no longer benefiting from treatment (disease progression or unacceptable toxicity had occurred), the participant withdrew consent, alternative access to study treatment was available and feasible, or until the end of the study, whichever occurred earlier.
- Arm B: Lenalidomide 20 mg (or 10 mg if CrCl Was 30 to <60 mL/Min) + Rituximab 375 mg/m^2: Participants received lenalidomide 20 mg (or 10 mg if creatinine clearance [CrCl] was 30 to less than [<] 60 milliliters per minute [mL/min]) capsule orally QD on Days 1 through 21 in each 28-day treatment cycle starting from Cycle 1 Day 1 until disease progression or unacceptable toxicity. Participants also received rituximab 375 mg/m^2 IV infusion on Day 1 of each 28-day treatment cycle from Cycles 1 to 6. After implementation of Protocol Amendment 1 (dated 08 June 2023), all participants were given the option either to continue with the randomized treatment arm or switch to ibrutinib monotherapy to receive ibrutinib 560 mg capsules orally QD until the investigator determined that the participant was no longer benefiting from treatment (disease progression or unacceptable toxicity had occurred), the participant withdrew consent, alternative access to study treatment was available and feasible, or until the end of the study, whichever occurred earlier.
Period: Overall Study
Arm/Group | Arm A1: Ibrutinib 560 mg + Rituximab 375 mg/m^2 | Arm A2: Ibrutinib 420 mg + Rituximab 375 mg/m^2 | Arm A3: Ibrutinib 140 mg + Rituximab 375 mg/m^2 | Arm B: Lenalidomide 20 mg (or 10 mg if CrCl Was 30 to <60 mL/Min) + Rituximab 375 mg/m^2
Started | 10 | 9 | 8 | 9
Participants Who Switched to Ibrutinib Monotherapy | 0 | 4 | 3 | 2
Completed | 10 | 9 | 8 | 8
Not Completed | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A1: Ibrutinib 560 mg + Rituximab 375 mg/m^2 | Arm A2: Ibrutinib 420 mg + Rituximab 375 mg/m^2 | Arm A3: Ibrutinib 140 mg + Rituximab 375 mg/m^2 | Arm B: Lenalidomide 20 mg (or 10 mg if CrCl Was 30 to <60 mL/Min) + Rituximab 375 mg/m^2 | Total
Number analyzed (Participants) | 10 | 9 | 8 | 9 | 36
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.5 (7.23) | 68.9 (8.08) | 64.6 (10.35) | 64.6 (7.60) | 66.2 (8.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 1 | 1 | 9
  Male | 6 | 6 | 7 | 8 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 2 | 3 | 10
  Not Hispanic or Latino | 7 | 7 | 6 | 6 | 26
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 2 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 2 | 4
  White | 6 | 7 | 4 | 5 | 22
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  BRAZIL | 5 | 2 | 2 | 3 | 12
  CZECH REPUBLIC | 0 | 0 | 1 | 0 | 1
  GREECE | 0 | 1 | 0 | 0 | 1
  MALAYSIA | 2 | 1 | 1 | 0 | 4
  POLAND | 1 | 1 | 0 | 2 | 4
  SPAIN | 1 | 1 | 1 | 0 | 3
  TAIWAN | 0 | 0 | 1 | 0 | 1
  THAILAND | 0 | 1 | 0 | 2 | 3
  TURKEY | 1 | 2 | 2 | 2 | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Leading to Discontinuation of Treatment: Arms A1, A2, A3 and B
Description: An adverse event (AE) was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs was defined as any new or worsening AE occurring at or after first dose of study treatment up to 30 days after last dose or prior to start of subsequent anticancer therapy, whichever occurred first. All TEAEs including serious and non-serious events were reported in this outcome measure.
Time Frame: From start of treatment (Day 1) up to 30 days after last dose of study drug or start of subsequent anticancer therapy, whichever occurred first (up to 12 months)
Population: Safety population was defined as all randomized participants of arms A1, A2, A3 and B who received at least 1 dose of any ibrutinib dosage level or control drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1: Ibrutinib 560 mg + Rituximab 375 mg/m^2 | Arm A2: Ibrutinib 420 mg + Rituximab 375 mg/m^2 | Arm A3: Ibrutinib 140 mg + Rituximab 375 mg/m^2 | Arm B: Lenalidomide 20 mg (or 10 mg if CrCl Was 30 to <60 mL/Min) + Rituximab 375 mg/m^2
Number analyzed (Participants) | 10 | 9 | 8 | 9
Participants
  Discontinuation of Treatment Ibrutinib/Lenalidomide | 1 | 0 | 0 | 2
  Discontinuation of Treatment Rituximab | 0 | 1 | 0 | 1

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Leading to Discontinuation of Treatment: Monotherapy Arm
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs was defined as any new or worsening AE occurring at or after first dose of study treatment up to 30 days after last dose or prior to start of subsequent anticancer therapy, whichever occurred first. All TEAEs included serious and non-serious events were reported in this outcome measure.
Time Frame: From start of monotherapy (post protocol amendment 1, dated 08 June 2023) up to 30 days after last dose of study drug or start of subsequent anticancer therapy, whichever occurred first (up to 6 months)
Population: Monotherapy population was defined as participants who were randomized to Arms A2, A3 and B and later switched to ibrutinib 560 mg QD monotherapy.
Measure: Count of Participants; unit: Participants
Groups:
- Monotherapy Arm: Ibrutinib 560 mg: Participants from Arm A2 (Ibrutinib 420 mg QD + Rituximab), Arm A3 (Ibrutinib 140 mg BID + Rituximab) and Arm B (Lenalidomide 20 mg + Rituximab) who were earlier receiving ibrutinib/lenalidomide + rituximab later switched to ibrutinib monotherapy post protocol amendment 1 (dated 08 June 2023), received ibrutinib 560 mg capsules orally QD (unless the dose was previously reduced) until the investigator determined that the participant was no longer benefiting from treatment (disease progression or unacceptable toxicity had occurred), the participant withdrew consent, alternative access to study treatment was available and feasible, or until the end of the study, whichever occurred earlier.
Arm/Group | Monotherapy Arm: Ibrutinib 560 mg
Number analyzed (Participants) | 9
Participants | 1

3. Primary Outcome: Number of Participants With Grade 3 or Higher TEAEs Based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version (v) 5.0: Arms A1, A2, A3 and B
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. TEAEs was defined as any new or worsening AE occurring at or after first dose of study treatment up to 30 days after last dose or prior to start of subsequent anticancer therapy, whichever occurred first. TEAEs were graded according to NCI-CTCAE v5.0 as Grade 1- Mild; Grade 2- Moderate; Grade 3- Severe or medically significant but not immediately life-threatening; Grade 4- Life-threatening consequences and Grade 5- Death related to AE. Number of participants with grade 3 or higher TEAEs (including serious and non-serious events) were reported in this outcome measure.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1: Ibrutinib 560 mg + Rituximab 375 mg/m^2 | Arm A2: Ibrutinib 420 mg + Rituximab 375 mg/m^2 | Arm A3: Ibrutinib 140 mg + Rituximab 375 mg/m^2 | Arm B: Lenalidomide 20 mg (or 10 mg if CrCl Was 30 to <60 mL/Min) + Rituximab 375 mg/m^2
Number analyzed (Participants) | 10 | 9 | 8 | 9
Participants | 7 | 3 | 5 | 8

4. Primary Outcome: Number of Participants With Grade 3 or Higher TEAEs Based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version (v) 5.0: Monotherapy Arm
Description: as for outcome 3
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy Arm: Ibrutinib 560 mg
Number analyzed (Participants) | 9
Participants | 1

5. Primary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (TESAEs): Arms A1, A2, A3 and B
Description: An AE was any untoward medical occurrence in a clinical study participant administered a medicinal (investigational or non-investigational) product. An AE does not necessarily have a causal relationship with the intervention. A serious AE was defined as any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a suspected transmission of any infectious agent via a medicinal product, or was medically important. TESAEs was defined as SAEs occurring at or after first dose of study treatment up to 30 days after last dose or prior to start of subsequent anticancer therapy, whichever occurred first.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1: Ibrutinib 560 mg + Rituximab 375 mg/m^2 | Arm A2: Ibrutinib 420 mg + Rituximab 375 mg/m^2 | Arm A3: Ibrutinib 140 mg + Rituximab 375 mg/m^2 | Arm B: Lenalidomide 20 mg (or 10 mg if CrCl Was 30 to <60 mL/Min) + Rituximab 375 mg/m^2
Number analyzed (Participants) | 10 | 9 | 8 | 9
Participants | 4 | 3 | 2 | 5

6. Primary Outcome: Number of Participants With Treatment Emergent Serious Adverse Events (TESAEs): Monotherapy Arm
Description: as for outcome 5
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy Arm: Ibrutinib 560 mg
Number analyzed (Participants) | 9
Participants | 1

7. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities: Hematology Parameters: Arms A1, A2, A3 and B
Description: Number of participants with clinical abnormalities in hematology laboratory parameters were reported. Hematology parameters included: Activated partial thromboplastin time (aPTT), hemoglobin, neutrophil count, white blood cell (WBC) count, lymphocyte count, platelet count and prothrombin international normalized ratio (INR). Abnormality criteria was assessed as per NCI CTCAE v5.0 grading, where Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening. Grade 0 was assigned when the laboratory value was not assigned a Grade 1 or higher. Only those categories in which at least 1 participant had data were reported.
Time Frame: From start of treatment (Day 1) up to 30 days after last dose of study drug (up to 12 months)
Population: Safety population was defined as all randomized participants of arms A1, A2, A3 and B who received at least 1 dose of any ibrutinib dosage level or control drug. Here, 'n' (number analyzed) signifies the participants analyzed for each specified parameter and n=0 signifies that there was no evaluable participant for specified parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1: Ibrutinib 560 mg + Rituximab 375 mg/m^2 | Arm A2: Ibrutinib 420 mg + Rituximab 375 mg/m^2 | Arm A3: Ibrutinib 140 mg + Rituximab 375 mg/m^2 | Arm B: Lenalidomide 20 mg (or 10 mg if CrCl Was 30 to <60 mL/Min) + Rituximab 375 mg/m^2
Number analyzed (Participants) | 10 | 9 | 8 | 9
Participants
  aPTT Prolonged Grade 1: number analyzed (Participants) | 1 | 0 | 0 | 0
  aPTT Prolonged Grade 1 | 1 |  |  |
  Hemoglobin Decreased Grade 0 | 3 | 2 | 2 | 0
  Hemoglobin Decreased Grade 1 | 3 | 6 | 4 | 5
  Hemoglobin Decreased Grade 2 | 3 | 1 | 1 | 1
  Hemoglobin Decreased Grade 3 | 1 | 0 | 1 | 3
  Hemoglobin Increased Grade 0 | 10 | 9 | 8 | 9
  Lymphocyte Count Decreased Grade 0 | 4 | 5 | 7 | 3
  Lymphocyte Count Decreased Grade 1 | 3 | 0 | 1 | 2
  Lymphocyte Count Decreased Grade 2 | 2 | 4 | 0 | 2
  Lymphocyte Count Decreased Grade 3 | 1 | 0 | 0 | 1
  Lymphocyte Count Decreased Grade 4 | 0 | 0 | 0 | 1
  Lymphocyte Count Increased Grade 0 | 8 | 8 | 7 | 6
  Lymphocyte Count Increased Grade 2 | 2 | 1 | 1 | 2
  Lymphocyte Count Increased Grade 3 | 0 | 0 | 0 | 1
  Neutrophil Count Decreased Grade 0 | 4 | 7 | 4 | 1
  Neutrophil Count Decreased Grade 1 | 1 | 1 | 0 | 1
  Neutrophil Count Decreased Grade 2 | 1 | 0 | 0 | 1
  Neutrophil Count Decreased Grade 3 | 2 | 1 | 4 | 2
  Neutrophil Count Decreased Grade 4 | 2 | 0 | 0 | 4
  Platelet Count Decreased Grade 0 | 2 | 2 | 5 | 1
  Platelet Count Decreased Grade 1 | 4 | 5 | 2 | 3
  Platelet Count Decreased Grade 2 | 2 | 1 | 0 | 3
  Platelet Count Decreased Grade 3 | 2 | 0 | 0 | 0
  Platelet Count Decreased Grade 4 | 0 | 1 | 1 | 2
  Prothrombin INR Increased Grade 0: number analyzed (Participants) | 1 | 0 | 0 | 0
  Prothrombin INR Increased Grade 0 | 1 |  |  |
  WBC Decreased Grade 0 | 3 | 4 | 5 | 3
  WBC Decreased Grade 1 | 5 | 5 | 3 | 2
  WBC Decreased Grade 2 | 1 | 0 | 0 | 3
  WBC Decreased Grade 3 | 1 | 0 | 0 | 0
  WBC Decreased Grade 4 | 0 | 0 | 0 | 1
  WBC Increased Grade 0 | 10 | 9 | 8 | 8
  WBC Increased Grade 3 | 0 | 0 | 0 | 1

8. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities: Hematology Parameters: Monotherapy Arm
Description: as for outcome 7
Time Frame: From start of monotherapy (post protocol amendment 1, dated 08 June 2023) up to 30 days after last dose of study drug (up to 6 months)
Population: Monotherapy population was defined as participants who were randomized to Arms A2, A3 and B and later switched to ibrutinib 560 mg QD monotherapy. Here 'N' (overall number of participants analyzed) refers to the number of participants evaluable for this outcome measure and 'n' (number analyzed) refers to number of participants analyzed for each specified parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy Arm: Ibrutinib 560 mg
Number analyzed (Participants) | 8
Participants
  aPTT Prolonged Grade 0: number analyzed (Participants) | 1
  aPTT Prolonged Grade 0 | 1
  Hemoglobin Increased Grade 0 | 8
  Hemoglobin Decreased Grade 0 | 2
  Hemoglobin Decreased Grade 1 | 5
  Hemoglobin Decreased Grade 2 | 1
  Lymphocyte Count Decreased Grade 0 | 5
  Lymphocyte Count Decreased Grade 1 | 1
  Lymphocyte Count Decreased Grade 2 | 1
  Lymphocyte Count Decreased Grade 4 | 1
  Lymphocyte Count Increased Grade 0 | 8
  Neutrophil Count Decreased Grade 0 | 6
  Neutrophil Count Decreased Grade 1 | 1
  Neutrophil Count Decreased Grade 2 | 1
  Platelet Count Decreased Grade 0 | 2
  Platelet Count Decreased Grade 1 | 6
  Prothrombin INR Increased Grade 0: number analyzed (Participants) | 1
  Prothrombin INR Increased Grade 0 | 1
  WBC Decreased Grade 0 | 5
  WBC Decreased Grade 1 | 3
  WBC Increased Grade 0 | 8

9. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities: Chemistry Parameters: Arms A1, A2, A3 and B
Description: Number of participants with clinical abnormalities in chemistry laboratory parameters were reported. Chemistry parameters included: sodium, aspartate aminotransferase (AST), potassium, alanine aminotransferase (ALT), creatinine, total bilirubin (BL), alkaline phosphatase, albumin, and calcium. Abnormality criteria was assessed as per NCI CTCAE v5.0 grading, where Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening. Grade 0 was assigned when the laboratory value was not assigned a Grade 1 or higher. Only those categories in which at least 1 participant had data were reported.
Time Frame: From start of treatment (Day 1) up to 30 days after last dose of study drug (up to 12 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A1: Ibrutinib 560 mg + Rituximab 375 mg/m^2 | Arm A2: Ibrutinib 420 mg + Rituximab 375 mg/m^2 | Arm A3: Ibrutinib 140 mg + Rituximab 375 mg/m^2 | Arm B: Lenalidomide 20 mg (or 10 mg if CrCl Was 30 to <60 mL/Min) + Rituximab 375 mg/m^2
Number analyzed (Participants) | 10 | 9 | 8 | 9
Participants
  ALT Increased Grade 0 | 5 | 9 | 8 | 6
  ALT Increased Grade 1 | 4 | 0 | 0 | 3
  ALT Increased Grade 3 | 1 | 0 | 0 | 0
  Albumin Decreased Grade 0 | 6 | 9 | 4 | 7
  Albumin Decreased Grade 1 | 2 | 0 | 4 | 1
  Albumin Decreased Grade 2 | 2 | 0 | 0 | 1
  Alkaline Phosphatase (AP) Increased Grade 0 | 8 | 8 | 5 | 7
  AP Increased Grade 1 | 2 | 1 | 3 | 2
  AST Increased Grade 0 | 5 | 8 | 8 | 6
  AST Increased Grade 1 | 4 | 1 | 0 | 3
  AST Increased Grade 3 | 1 | 0 | 0 | 0
  Bilirubin (BL) Increased Grade 0 | 7 | 7 | 7 | 8
  BL Increased Grade 1 | 2 | 2 | 0 | 1
  BL Increased Grade 2 | 0 | 0 | 1 | 0
  BL Increased Grade 3 | 1 | 0 | 0 | 0
  Calcium Corrected Decreased Grade 0 | 7 | 7 | 6 | 6
  Calcium Corrected Decreased Grade 1 | 3 | 2 | 2 | 2
  Calcium Corrected Decreased Grade 2 | 0 | 0 | 0 | 1
  Calcium Corrected Increased Grade 0 | 10 | 9 | 8 | 8
  Calcium Corrected Increased Grade 1 | 0 | 0 | 0 | 1
  Creatinine Increased Grade 0 | 9 | 7 | 4 | 6
  Creatinine Increased Grade 1 | 1 | 2 | 2 | 3
  Creatinine Increased Grade 2 | 0 | 0 | 2 | 0
  Potassium Decreased Grade 0 | 7 | 7 | 6 | 9
  Potassium Decreased Grade 2 | 2 | 1 | 2 | 0
  Potassium Decreased Grade 4 | 1 | 1 | 0 | 0
  Potassium Increased Grade 0 | 10 | 8 | 7 | 9
  Potassium Increased Grade 2 | 0 | 1 | 1 | 0
  Sodium Decreased Grade 0 | 7 | 6 | 5 | 8
  Sodium Decreased Grade 1 | 3 | 3 | 3 | 1
  Sodium Increased Grade 0 | 8 | 9 | 8 | 8
  Sodium Increased Grade 1 | 2 | 0 | 0 | 1

10. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities: Chemistry Parameters: Monotherapy Arm
Description: Number of participants with clinical abnormalities in chemistry laboratory parameters were reported. Chemistry parameters included: sodium, aspartate aminotransferase (AST), potassium, alanine aminotransferase (ALT), creatinine, total bilirubin, alkaline phosphatase, albumin, and calcium. Abnormality criteria was assessed as per NCI CTCAE v5.0 grading, where Grade 1 = mild; Grade 2 = moderate; Grade 3 = severe; Grade 4 = life-threatening. Grade 0 was assigned when the laboratory value was not assigned a Grade 1 or higher. Only those categories in which at least 1 participant had data were reported.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Monotherapy Arm: Ibrutinib 560 mg
Number analyzed (Participants) | 8
Participants
  ALT Increased Grade 0 | 8
  Albumin Decreased Grade 0 | 6
  Albumin Decreased Grade 1 | 2
  Alkaline Phosphatase Increased Grade 0 | 8
  AST Increased Grade 0 | 8
  Bilirubin Increased Grade 0 | 8
  Calcium Corrected Decreased Grade 0 | 7
  Calcium Corrected Decreased Grade 1 | 1
  Calcium Corrected Increased Grade 0 | 8
  Creatinine Increased Grade 0 | 7
  Creatinine Increased Grade 1 | 1
  Potassium Decreased Grade 0 | 7
  Potassium Decreased Grade 2 | 1
  Potassium Increased Grade 0 | 8
  Sodium Decreased Grade 0 | 5
  Sodium Decreased Grade 1 | 3
  Sodium Increased Grade 0 | 8

ADVERSE EVENTS:
Time Frame: Arm A1, A2, A3 and B: From start of treatment (Day 1) up to 30 days after last dose of study drug or start of subsequent anticancer therapy, whichever occurred first (up to 12 months); Monotherapy arm: From start of monotherapy (post protocol amendment 1, dated 08 June 2023) up to 30 days after last dose of study drug or start of subsequent anticancer therapy, whichever occurred first (up to 6 months)
Description: Arm A1, A2, A3 and B: Safety population was defined as all randomized participants of arms A1, A2, A3 and B who received at least 1 dose of any ibrutinib dosage level or control drug. Monotherapy population was defined as participants who were randomized to Arms A2, A3 and B and later switched to ibrutinib 560 mg QD monotherapy.
Arm/Group | Arm A1: Ibrutinib 560 mg + Rituximab 375 mg/m^2 | Arm A2: Ibrutinib 420 mg + Rituximab 375 mg/m^2 | Arm A3: Ibrutinib 140 mg + Rituximab 375 mg/m^2 | Arm B: Lenalidomide 20 mg (or 10 mg if CrCl Was 30 to <60 mL/Min) + Rituximab 375 mg/m^2 | Monotherapy Arm: Ibrutinib 560 mg
All-Cause Mortality (participants affected / at risk) | 1/10 | 0/9 | 1/8 | 2/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 4/10 | 3/9 | 2/8 | 5/9 | 1/9
Other Adverse Events (participants affected / at risk) | 10/10 | 7/9 | 8/8 | 8/9 | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A1: Ibrutinib 560 mg + Rituximab 375 mg/m^2 (N=10) | Arm A2: Ibrutinib 420 mg + Rituximab 375 mg/m^2 (N=9) | Arm A3: Ibrutinib 140 mg + Rituximab 375 mg/m^2 (N=8) | Arm B: Lenalidomide 20 mg (or 10 mg if CrCl Was 30 to <60 mL/Min) + Rituximab 375 mg/m^2 (N=9) | Monotherapy Arm: Ibrutinib 560 mg (N=9)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Septic Shock (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Skin Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Adenocarcinoma Metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Cerebellar Haemorrhage (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Hypertensive Crisis (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A1: Ibrutinib 560 mg + Rituximab 375 mg/m^2 (N=10) | Arm A2: Ibrutinib 420 mg + Rituximab 375 mg/m^2 (N=9) | Arm A3: Ibrutinib 140 mg + Rituximab 375 mg/m^2 (N=8) | Arm B: Lenalidomide 20 mg (or 10 mg if CrCl Was 30 to <60 mL/Min) + Rituximab 375 mg/m^2 (N=9) | Monotherapy Arm: Ibrutinib 560 mg (N=9)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 3 | 0
Eosinophilia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 4 | 1 | 4 | 4 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 3 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Cardiac Failure (Cardiac disorders) | 0 | 0 | 1 | 0 | 1
Conjunctivitis Allergic (Eye disorders) | 1 | 0 | 0 | 0 | 0
Ocular Hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 1
Periorbital Oedema (Eye disorders) | 0 | 0 | 2 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 3 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1 | 0
Odynophagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0
Extravasation (General disorders) | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0 | 0
Infusion Site Rash (General disorders) | 0 | 0 | 0 | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0 | 1 | 1 | 0
Puncture Site Haematoma (General disorders) | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 0
Anaphylactic Reaction (Immune system disorders) | 0 | 0 | 1 | 0 | 0
Body Tinea (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0
Fungal Foot Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Herpes Zoster (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Oral Herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 1 | 0 | 0
Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Skin Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Soft Tissue Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1 | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Infusion Related Reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 1 | 0 | 1 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 2 | 0 | 0
Blood Immunoglobulin M Decreased (Investigations) | 0 | 1 | 0 | 0 | 0
Blood Lactate Dehydrogenase Decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood Lactate Dehydrogenase Increased (Investigations) | 0 | 0 | 0 | 1 | 0
Hepatic Enzyme Increased (Investigations) | 1 | 0 | 0 | 0 | 0
Neutrophil Count Decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Neutrophil Count Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Platelet Count Decreased (Investigations) | 0 | 0 | 2 | 2 | 0
Platelet Count Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Weight Decreased (Investigations) | 0 | 1 | 0 | 0 | 0
White Blood Cell Count Increased (Investigations) | 0 | 0 | 1 | 0 | 0
Glucose Tolerance Impaired (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1
Iron Deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Meningioma Benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Ischaemic Stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Renal Impairment (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0
Epiglottic Cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Oropharyngeal Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Nail Bed Inflammation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1 | 0
Purpura (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Aortic Dilatation (Vascular disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 5 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-06-08): https://cdn.clinicaltrials.gov/large-docs/52/NCT05564052/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/52/NCT05564052/SAP_002.pdf